CLINICAL TRIAL: NCT05891691
Title: THE EFFECTS OF A PROGRAM OF MOVING MUSIC ACTIVITIES, YOGA AND MASSAGE ON HEALTHY PRESCHOOL CHILDREN'S SOCIAL EMOTIONAL WELL-BEING AND PSYCHOLOGICAL RESILIENCE, SOCIAL SKILLS AND QUALITY OF LIFE
Brief Title: THE EFFECTS OF THE YOGA-BASED PROGRAM ON THE SOCIAL EMOTIONAL AND PSYCHOLOGICAL HEALTH OF CHILDREN, SOCIAL SKILLS AND QUALITY OF LIFE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Gökçe Algül, lecturer, Gazi University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Gazi University-GokceAlgul-001
Record Dates: First submitted 2023-05-18; First posted 2023-06-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-05

CONDITIONS: Preschool; Yoga; Massage; Psychological Well-Being; Quality of Life
MeSH Terms: conditions — Psychological Well-Being | interventions — Yoga; Massage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): In addition to the training program prepared by the classroom teacher, the initiative group will receive a program that includes music activities, yoga postures accompanied by stories, breathing techniques and massage exercises, 2 days a week, 30 minutes a day for 6 weeks.
  Interventions: Behavioral: Music Activities, Yoga, Massage
- Control Group (No Intervention): The teachers will continue their education within the program they have prepared.

INTERVENTIONS:
Behavioral: Music Activities, Yoga, Massage — The program begins with music and dance movements using percussion instruments (rhythm stick, stone triangle, drum, cymbal, tambourine, maracas, etc.) and body percussion. In this phase, the children will follow the instructions of the researcher. The goal is to warm up the bodies and musically experience the beginning of the program After the warm-up, yoga postures are combined with breathing techniques that focus on developing awareness of body sensations and feelings.The daily program ends with massage. During the massage application, the children sit in a circle. The massage is performed by the children observing the movements of the researcher on their arms and legs and applying them on their own arms and legs.Yoga postures, breathing techniques, and massage practices are accompanied by stories to ensure children's active participation, encourage their development, and facilitate their acquisition of new approaches.
  Arms: Intervention Group

SUMMARY:
This study was planned to evaluate the effectiveness of a yoga-based psychosocial development program developed in line with the literature to improve the social, emotional and behavioral skills and quality of life of healthy preschool children. Watson's Human Care Model constitutes the theoretical framework of the study. The sample of the study, which will be conducted in a quasi-experimental design with a pre-test-post-test control group, consists of healthy children aged 60-72 months. The g*power 3.1.9.4 program was used to determine the sample size and it was determined that there should be at least 34 people in each group. The program consists of moving music activities, yoga postures accompanied by stories, breathing techniques and self-massage practices. The program will be implemented by the researcher, who has received specialty training in child yoga, for 30 minutes a day, two days a week for 6 weeks. Data will be collected using the Parent and Child Descriptive Data Form, Program Participation Form, Child Self-Assessment Form, Social Emotional Well-Being and Psychological Resilience Scale for Preschool Children, Social Competence and Behavior Rating Scale-30 and Pediatric Quality of Life Inventory. As a result of this study, positive effects are expected on the social, emotional, behavioral skills and quality of life of children to whom the psychosocial development program is applied.

DETAILED DESCRIPTION:
Preschool years are a critical period in which children acquire physical, mental, emotional and social skills and development progresses rapidly. Psychosocial skills are one of the most important dimensions of development. It is emphasized that there is an important relationship between psychosocial skills and health and well-being. It is reported that socially competent and social-emotionally developed children are better able to cope with stressful situations, this skill increases school readiness, academic self-efficacy and academic success, and improves peer relations and coping skills with emotions. In the literature, school-based intervention programs that facilitate children's coping with stress, enable them to respond constructively to psychological and social difficulties, and help them develop emotion regulation skills are recommended from preschool onwards. The aim of this study was to determine the effects of a psychosocial development program that includes moving music activities, exercises including yoga postures accompanied by stories, breathing techniques and self-massage practices on social-emotional well-being and psychological resilience, social competence, behavior and quality of life of preschool children.

ELIGIBILITY:
Inclusion Criteria:

* 60-72 months
* Do not have a health problem that would prevent them from actively participating in group games (attention deficit, hyperactivity, down syndrome, autism, etc.)
* Who have not participated in a similar program before
* Speak and understand Turkish
* Volunteer to participate in the program
* Children whose parents gave consent to participate in the study.

Exclusion Criteria:

* She has a contraindication such as heart disease, wilms tumor that would prevent her from doing massage and yoga

Ages: 60 Months to 72 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 68 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Social Emotional Wellbeing and Psychological Resilience Scale for Preschool Children | Baseline, after the six week intervention.
  A 36 item scale validated with six sub-scales: Communicating / Social Performance, Self-Control / Thoughtfulness, Assertiveness, Emotional Stability / Coping with Stress, Task Orientation, Enjoyment of Exploration. The scale will be completed by teachers on behalf of the children to screen and monitor the response to the intervention.
Social Competence and Behavior Evaluation SCBE-30 | Baseline, after the six week intervention.
  A 30 item scale validated with three sub-scales: Competence, Anger-Aggression, and Anxiety-Introversion, with ten items in each dimension.The scale will be completed by teachers on behalf of the children to screen and monitor the response to the intervention.
The Pediatric Quality of Life Inventory (PedsQL) (5-7 years) | Baseline, after the six week intervention.
  It consists of 23 items questioning physical and psychosocial (emotional, social and school functionality) functionality. The scale will be completed by parents on behalf of the children to screen and monitor the response to the intervention.

SECONDARY OUTCOMES:
Qualitative Data on the Feasibility of Yoga Intervention Using Focus Group Discussions with Children | After six weeks
  At the end of 6 weeks, a semi-structured qualitative interview will be conducted with a simple random method with 10 randomly selected children from the intervention group to evaluate the program. Children will be asked what they liked most and least about the program, what they learned from yoga, their favorite poses in yoga, how breathing exercises felt. Interviews with the children will be held in a quiet, uninterrupted, school-owned area to be directed by the school administration. In order for the children to feel more comfortable, the children will be interviewed in groups of two or three.
Program Attendance Form | During the six-week intervention, before yoga-based practice classes
  Will assess the number of school-based sessions each child attends to assess commitment to the program.
Self-Assessment Form for Children | During the six-week intervention, after yoga-based practice classes
  A visual analog scale will be used to measure each child's satisfaction and comfort levels in the intervention group.
Parent and Child Descriptive Data Form | Baseline
  A total of 12 questions (age, sex, education level, monthly income, etc.) were asked about the child and parent's identifying information. The descriptive characteristics form was developed by the researchers based on the literature